CLINICAL TRIAL: NCT05329584
Title: An Assessment of Two Accelerated Rehabilitation Programs for Use With the InSpaceTM Subacromial Tissue Spacer System in the Treatment of Full-thickness Massive, Irreparable Rotator Cuff Tears
Brief Title: InSpace Accelerated Rehabilitation Study
Acronym: iAccelerate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Endoscopy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYK-SM-2021-01
Record Dates: First submitted 2022-03-17; First posted 2022-04-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group I (Experimental): InSpace device + accelerated rehabilitation in a formalized program (FP)
  Interventions: Device: InSpace Subacromial Tissue Spacer
- Group II (Experimental): InSpace device + accelerated rehabilitation in an at-home program (AHP)
  Interventions: Device: InSpace Subacromial Tissue Spacer

INTERVENTIONS:
Device: InSpace Subacromial Tissue Spacer — Rotator Cuff Tear Treatment

SUMMARY:
This is a prospective, parallel group, open-label, multi- center, randomized study to assess two accelerated rehabilitation programs for use with the InSpace device in the treatment of full thickness Massive, Irreparable Rotator Cuff Tears (MIRCTs) performed during an arthroscopic procedure.

DETAILED DESCRIPTION:
Study Objectives:

Primary:

• To evaluate clinical outcomes of both a formalized or an at-home rehabilitation program when used in conjunction with the InSpace device as compared to the corresponding InSpace Pivotal study results.

* To demonstrate consistency of each intervention group with the corresponding historical control study results.
* To demonstrate that comparable clinical outcomes can be achieved for each intervention group.

Secondary:

• Change in clinical outcomes compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST meet ALL the following criteria to be included in the study:

* The subject has signed the IRB approved Informed Consent Form (ICF) specific to this study prior to enrollment
* Is male or female ≥ sixty-five (65) years of age
* Positive diagnostic imaging by MRI within 9 months of enrollment of the index shoulder indicating a full thickness MRCT:

  * Measuring ≥ 5 cm in diameter
  * Involving ≥ two tendons
* Functional deltoid muscle and preserved passive range of motion on physical examination
* Documented VAS score > 30 mm pain
* Failed non-operative treatment of at least 3 months from the initial treatment to include one or more of the following:

  * Oral analgesics
  * Anti-inflammatory medication (e.g., ibuprofen, naproxen)
  * Corticosteroid injection(s)
  * Physical therapy
  * Activity modification
  * Rest (sling used)
* Must be able to read and understand the approved Informed Consent Form (written and oral)
* Must be in general good health (as determined by the Investigator) based on screening assessments and medical history
* Must be independent, ambulatory, and can comply with all post-operative evaluations, visits, and electronic database collection

Intra-operative Inclusion Criteria

Subjects MUST meet the following criteria to be randomized in the study:

* Full thickness tear
* Tear size ≥ 5 cm in diameter
* Tear involving ≥ two tendons

Exclusion Criteria:

Subjects will be excluded from the study, if they meet ANY of the following individual exclusion criteria:

* Known allergy to the device material (copolymer of PLA (poly (lactic acid) and -ε-caprolactone)
* Evidence of the following conditions:

  * Severe gleno-humeral or acromio-humeral arthritis
  * Full thickness cartilage loss as seen on MRI
  * History within the past 5 years of anterior or posterior shoulder subluxation or dislocation as determined by history, examination, or radiographic findings
  * Pre-existing deltoid defect or deltoid palsy
  * Major joint trauma, infection, or necrosis
  * Partial thickness tears of the supraspinatus
  * Fully reparable rotator cuff tear [Tear of less than 5 cm in diameter (or < 4 cm2) with retractable tendon that can be fully repaired]
  * Known neurovascular compromise
  * Complete deltoid muscle palsy
  * Traumatic muscle tears of the pectoralis or deltoid
* The subject requires concomitant:

  * Subscapularis repair
  * Labral repair of any type
  * Biceps tenodesis
* Previous surgery of the index shoulder in the past 1 year, excluding diagnostic arthroscopy
* The subject's condition is bilateral and rotator cuff repair is scheduled or to be scheduled over the course of this study for the contra lateral shoulder
* Major medical condition that could affect quality of life and influence the results of the study (e.g., rheumatoid arthritis)
* The subject has documented evidence of a history (e.g., liver testing) of drug/alcohol abuse within 12 months of enrollment
* The subject's condition represents a worker's compensation case
* The subject is currently involved in a health-related litigation procedure
* Females of child-bearing potential who are pregnant or plan to become pregnant.
* Concurrent participation in an investigational clinical study one month prior to enrollment or during the entire study period
* The subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.), to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant to follow-up
* The subject is receiving prescription narcotic pain medication for conditions unrelated to the index shoulder condition
* The subject currently has an acute infection in the area surrounding the surgical site.
* Baseline WORC score less than 420

Intra-operative Exclusion Criteria:

Subjects will not be randomized and will be terminated from the study if they meet ANY of the following individual intra-operative exclusion criteria:

* Rotator cuff is/presents with:

  * Fully reparable with adequate tissue and muscle quality (equivalent to Goutallier stage 1 or 2)
  * Partial thickness tear of the supraspinatus
  * Evidence of significant osteoarthritis
* The subject requires concomitant:

  * Subscapularis repair
  * Labral repair of any type
  * Biceps tenodesis
* Coracoacromial ligament functional deficiency or shoulder instability is identified

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in American Shoulder and Elbow (ASES) Score | Day 0 through Month 12
  This is a subject self-report questionnaire and Investigator assessment questionnaire. The subject portion collects information on activities of daily living (i.e., 10 questions). The Investigator assessment portion documents ROM (forward elevation/flexion, external rotation, internal rotation, cross-body adduction), signs, strength, and instability. ASES minimal clinical important difference (MCID) and substantial clinical benefit (SCB) have been previously described for the ASES score in patients undergoing rotator cuff repair as 11.1 and 17.5, respectively.
  Change in American Shoulder and Elbow Surgeons (ASES) Score will be expressed as the percentages demonstrating a minimal clinical important difference (MCID; ASES ≥ 11.1) and the substantial clinical benefit (SCB; ASES ≥ 17.5) in ASES from baseline at Month 12. Minimum value: 0, Maximum value: 100 (with a higher score indicating a better outcome).

SECONDARY OUTCOMES:
Safety Assessment | Day 0 through Month 24
  • Safety will be evaluated by type, frequency, severity, and relatedness of adverse events to study intervention at each follow-up visit through Month 24
Change in Western Ontario Rotator Cuff (WORC) Score | Day 0 through Month 24
  Change in WORC Score from baseline. Minimum value: 2,100, Maximum value: 0 (with a lower score indicating a better outcome).
  This is a subject self-report questionnaire that is a disease-specific Quality of Life Measurement Tool specifically designed to evaluate quality of life in persons with pathology of the rotator cuff. It is comprised of 21 items in 5 domains (i.e., physical symptoms, sports and recreation, work, lifestyle, emotions).
Change in Constant Score (CS) Outcome Score | Day 0 through Month 24
  Change in CS Outcome Score from baseline. Minimum value: 0, Maximum value: 100 (with a higher score indicating a better outcome).
  This is a self-reported questions as well as Investigator or designee performed assessment of the shoulder. The tool is divided into four subscales: pain, activities of daily living, strength and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder.
Change in EuroQol 5-Dimensions Questionnaire (EQ-5D-5L) Score | Day 0 through Month 24
  Change in EQ-5D-5L Score from baseline. Minimum value: 0, Maximum value: 100 (with a higher score indicating a better outcome).
  This is a subject self-report questionnaire to measure health-related quality of life (HRQOL). It consists of 5 questions capturing the subject's current health across five dimensions (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). It also includes a numerical visual analogue scale (EQ-VAS).
Change in Visual Analog Scale (VAS) Score | Day 0 through Month 24
  Change in VAS Score from baseline. This is a subject self-report questionnaire to measure pain. The patient marks on the line the point that they feel represents their perception of their current state. The amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. (An extreme amount of pain would be considered a worse outcome)
Change in Range of Motion (ROM) Score | Day 0 through Month 24
  Change in ROM Score from baseline. Minimum value: 0, Maximum value: 180 (with a higher score indicating a better outcome).
Change in Single Assessment Numeric Evaluation (SANE) Score | Day 0 through Month 24
  Change in SANE from baseline. Minimum value: 0%, Maximum value: 100% (with 100% being normal).
  This is a subject self-report questionnaire to measure function. The patient marks on the line the point that they feel represents their perception of their current state of functional improvement. Example: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
Patient's satisfaction with their procedure | Month 12 and Month 24
  Patient Satisfaction Score at Month 12 and Month 24.
  This is a single-question to evaluate the patients' current state of satisfaction. Responses are binary with Yes or No answers. ('Yes' would be considered a positive outcome)
Costing | Day 0 through Month 24
  Costs associated with all visits
Time to Recovery | Day 0 through Month 24
  Time to recovery by cumulative time between discharge and return to driving
Analgesia Use | Day 0 through Month 24
  Analgesia use (drug and frequency)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Roden, MS, Study Director — Stryker Endoscopy
Locations (11):
- United States (11):
  - Musculoskeletal-Orthopedic Research and Education Foundation, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Steadman Hawkins Clinic Denver, Englewood, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Paley Orthopaedics & Spine, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - The Rothman Institute, Philadelphia, Pennsylvania
  - TSAOG Orthopaedics & Spine, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No